CLINICAL TRIAL: NCT05955768
Title: Clinical Study on "Pain Control of Cervical Dilation by Lidocaine Solution Injected Into a Single-use Micro-non-invasive Injection Cervical Dilator"
Brief Title: Clinical Study on "Pain Control of Cervical Dilation by Lidocaine Solution Injected Into a Disposable Cervical Dilator"
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023001
Record Dates: First submitted 2023-07-04; First posted 2023-07-21 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-06

CONDITIONS: Cervical Dilatations
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial group (Experimental): Disposable cervical dilator stick combined with lidocaine hydrochloride injection.
  Interventions: Procedure: Disposable cervical dilator stick combined with lidocaine hydrochloride injection
- Control group (Placebo Comparator): Disposable cervical dilator stick combined with normal saline injection.
  Interventions: Procedure: Disposable cervical dilator stick combined with normal saline injection

INTERVENTIONS:
Procedure: Disposable cervical dilator stick combined with lidocaine hydrochloride injection — The subject will undergo routine disinfection and receive cervical paracervical nerve block anesthesia (5mL of 1% lidocaine injection at the level of the bilateral sacral ligaments). After waiting for 2 minutes, the researcher gently checks the depth of the uterine cavity with a probe and then remove it. The nurse connects the disposable cervical dilator to the syringe containing lidocaine hydrochloride. The researcher inserts the disposable cervical dilator into the cervical canal in line with the probe direction, and slowly inject drug from the syringe into it within a minute. The researcher waits for another minute before removing the disposable cervical dilator. The researcher removes the IUD with a ring hook. If necessary, the researcher will use metal Hegar dilators to dilate cervix.
  Arms: Trial group
Procedure: Disposable cervical dilator stick combined with normal saline injection — The subject will undergo routine disinfection and receive cervical paracervical nerve block anesthesia (5mL of 1% lidocaine injection at the level of the bilateral sacral ligaments). After waiting for 2 minutes, the researcher gently checks the depth of the uterine cavity with a probe and then remove it. The nurse connects the disposable cervical dilator to the syringe containing normal saline. The researcher inserts the disposable cervical dilator into the cervical canal in line with the probe direction, and slowly inject drug from the syringe into it within a minute. The researcher waits for another minute before removing the disposable cervical dilator. The researcher removes the IUD with a ring hook. If necessary, the researcher will use metal Hegar dilators to dilate cervix.
  Arms: Control group

SUMMARY:
This study is a multicenter, randomized (each group was assigned 1:1), double-blind controlled trial.

This study aims to investigate if lidocaine injection into the single-use micro-non-invasive injection cervical dilator (short for disposable cervical dilators) leads to better pain control efficacy compared with normal saline injection in intrauterine device(short for IUD) removal surgery. Furthermore, this study aims to compare cervical dilation degree, safety, and patient satisfaction between groups.

Research objects Between August 1, 2023, and August 1, 2025, 74 healthy women who voluntarily request the removal of the intrauterine device under local anesthesia in Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine.

The subjects will be dividied into two groups at random.

1. Trial group: disposable cervical dilator stick combined with lidocaine hydrochloride injection.
2. Control group: disposable cervical dilator stick combined with normal saline injection.

Intervention measures:

The nurse fill the syringe with 5ml of either 2% lidocaine hydrochloride injection or normal saline based on the group allocation specified. The appearance of the two drugs is indistinguishable after loading.

The subject will undergo routine disinfection and receive cervical paracervical nerve block anesthesia. After waiting for 2 minutes, the researcher gently checks the depth of the uterine cavity with a probe and then remove it. After that, the researcher tries to insert a number 10 to 4 metal Hegar dilator in sequence, until passes through the internal cervical orifice without resistance. The nurse connects the disposable cervical dilator to the syringe containing drug. The researcher inserts the disposable cervical dilator into the cervical canal in line with the probe direction, and slowly inject drug from the syringe into it within a minute. The researcher waits for another minute before removing the disposable cervical dilator. After that, the researcher tries to insert a number 10 to 4 metal Hegar dilator in sequence, until passes through the internal cervical orifice without resistance.

The researcher removes the IUD with a ring hook. If necessary, the researcher will use metal Hegar dilators to dilate cervi. The subject uses VAS to evaluate the degree of pain before, during and after surgery. Oral antibiotics were routinely given post-surgery to prevent infection.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and <65 years old;
2. Voluntary request for removal of intrauterine device under local anesthesia;
3. No known allergic reactions or sensitivity to lidocaine, physiological saline and polyvinyl formaldehyde polymer materials in the past;
4. Volunteer participation in this study.

Exclusion Criteria:

1. Dysplasia of uterine cavity structure;
2. Known lesions such as uterine fibroids that compress and cause uterine cavity deformation;
3. Presence of untreated acute cervicitis or pelvic inflammatory diseases;
4. History of cervical surgery;
5. Systemic diseases that can affect pain perception;
6. Current or past use of illegal drugs or anesthetic and analgesic drugs;
7. Unable to understand how to score pain using Visual Analog Scale (short for VAS).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) pain score | Baseline
  The subject uses VAS to evaluate the degree of pain before surgery. Visual analog scale pain score (VAS score), minimum 0mm, maximum 100mm, higher value means more severe pain.
Visual analog scale (VAS) pain score | Intraoperative
  The subject uses VAS to evaluate the degree of pain at the most painful time during the surgery. Visual analog scale pain score (VAS score), minimum 0mm, maximum 100mm, higher value means more severe pain.
Visual analog scale (VAS) pain score | 30 minutes after surgery
  The subject uses VAS to evaluate the degree of pain 30 minutes after surgery. Visual analog scale pain score (VAS score), minimum 0mm, maximum 100mm, higher value means more severe pain.

SECONDARY OUTCOMES:
Cervical dilatation | Baseline
  Before dilation, the researcher tries to insert a number 10 to 4 metal Hegar dilator in sequence, until passes through the internal cervical orifice without resistance. The researcher records the diameter of the last dilator as the predilated cervical dilation score. The minimum value of cervical dilation is 4, and the maximum value is 10. If the actual dilation of the cervix is not within the measurement range, it is recorded as less than 4 or greater than 10. The larger the value, the greater the degree of cervical dilation.
Cervical dilatation | Within one minute after using the disposable cervical dilator
  Within one minute after using the disposable cervical dilator, the researcher tries to insert a number 10 to 4 metal Hegar dilator in sequence, until passes through the internal cervical orifice without resistance. The researcher records the diameter of the last dilator as the postdilated cervical dilation score. The minimum value of cervical dilation is 4, and the maximum value is 10. If the actual dilation of the cervix is not within the measurement range, it is recorded as less than 4 or greater than 10. The larger the value, the greater the degree of cervical dilation.

CONTACTS AND LOCATIONS:
Overall Officials: Yahui Yahui, Yahui, Principal Investigator — Zhejiang University
Locations (1):
- Hangzhou First People's Hospita, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
If necessary, other researchers can ask us to share the raw data via email after the results are published.

REFERENCES:
- [Background] Aksoy H, Aksoy U, Ozyurt S, Acmaz G, Babayigit M. Lidocaine 10% spray to the cervix reduces pain during intrauterine device insertion: a double-blind randomised controlled trial. J Fam Plann Reprod Health Care. 2016 Apr;42(2):83-7. doi: 10.1136/jfprhc-2014-100917. Epub 2015 Mar 10. PMID 25759418
- [Background] Falcone F, Raimondo G, Stark M, Dessole S, Torella M, Raimondo I. Balloon Catheter for Cervical Priming before Operative Hysteroscopy in Young Women: A Pilot Study. J Invest Surg. 2020 Apr;33(4):301-306. doi: 10.1080/08941939.2018.1503379. Epub 2018 Oct 31. PMID 30380354
- [Background] Charoenkwan K, Nantasupha C. Methods of pain control during endometrial biopsy: A systematic review and meta-analysis of randomized controlled trials. J Obstet Gynaecol Res. 2020 Jan;46(1):9-30. doi: 10.1111/jog.14152. Epub 2019 Oct 30. PMID 31667985
- [Background] Babandi RM, Agboghoroma OC, Durojaiye KW, Jimoh KO, Essiet EA. Pain Relief for Hysterosalpingography: A Randomized Controlled, Double Blinded Trial Comparing Suppository Diclofenac, Prilocaine/Lignocaine (EMLA) Cream And Placebo. West Afr J Med. 2021 Dec 30;38(12):1174-1182. PMID 35035229
- [Background] Abbas AM, Abdellah MS, Khalaf M, Bahloul M, Abdellah NH, Ali MK, Abdelmagied AM. Effect of cervical lidocaine-prilocaine cream on pain perception during copper T380A intrauterine device insertion among parous women: A randomized double-blind controlled trial. Contraception. 2017 Mar;95(3):251-256. doi: 10.1016/j.contraception.2016.10.011. Epub 2016 Nov 4. PMID 27823944
- [Result] Veces A, Reyes O. Use of Topical Lidocaine Gel Plus Paracervical Blockade vs. Paracervical Blockade Alone for Pain Management During Manual Vacuum Aspiration: ADouble-Blind, Randomized, Placebo-Controlled Trial. J Obstet Gynaecol Can. 2019 May;41(5):641-646. doi: 10.1016/j.jogc.2018.05.027. Epub 2018 Oct 26. PMID 31007170